CLINICAL TRIAL: NCT02334358
Title: A Multi-center, Prospective and Observational Study to Evaluate Long-term Safety and Biodegradability of YVOIRE Classic s Injected Into the Nasolabial Folds
Brief Title: Observational Study to Evaluate Long-term Safety and Biodegradability of YVOIRE Classic s
Status: Completed | Type: Observational
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-HAOS004
Record Dates: First submitted 2015-01-04; First posted 2015-01-08 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2018-11

CONDITIONS: Correction of Nasolabial Folds

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- YVOIRE Classic s: Treatment with YVOIRE Classic s
  Interventions: Device: YVOIRE Classic s

INTERVENTIONS:
Device: YVOIRE Classic s

SUMMARY:
To evaluate long-term safety of YVOIRE classic s by incidence of adverse events including injection site local reactions and biodegradability

ELIGIBILITY:
Inclusion Criteria:

1. Subjects whose age is over 18 years old
2. Subjects whose WSRS grade is equal or greater than 2
3. Subjects must be willing and able to provide written informed consent
4. Subjects who are scheduled to be treated with YVOIRE classic s for facial tissue augmentation to correct the nasolabial folds

Exclusion Criteria:

1. Subjects who are sensitive to hyaluronic acid or any excipients of YVOIRE classic s
2. Subjects who have received permanent implantation (silicone, PAAG, PMMA, CaHA etc) on the nasolabial folds
3. Subjects who have received nonpermanent aesthetic treatments, such as botulinum toxin injection or filler on the nasolabial folds within 9 months before screening
4. Subjects who have received face lifting or plastic surgery on face within 9 months before screening
5. Subjects who have received laser therapy on the nasolabial folds, chemical peeling or peeling on face within 3 months before the screening
6. Subjects who have any skin diseases (including inflammation and skin cancer) or infectious diseases on the injection sites
7. Subjects who tend to have hypertrophic scars
8. Subjects with a history of streptococcal disease, severe allergy or anaphylaxis or bleeding disorders.
9. Women in pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject who receive hyaluronic acid filler into the nasolabial folds
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Q Li, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China

RESULTS

PARTICIPANT FLOW:
Groups:
- YVOIRE Classic s: YVOIRE Classic s
Period: Overall Study
Arm/Group | YVOIRE Classic s
Started | 503
Completed | 494
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | YVOIRE Classic s
Number analyzed (Participants) | 494
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.44 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 480
  Male | 14
Region of Enrollment [Number; unit: participants]
  China | 494

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Device-related Adverse Events
Time Frame: Until subject reaching total biodegradation criterion (WSRS change) ; an expected average of 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | YVOIRE Classic s
Number analyzed (Participants) | 503
Participants | 16

ADVERSE EVENTS:
Time Frame: Until subject reaching total biodegradation criterion (WSRS change) ; an expected average of 2 years.
Arm/Group | YVOIRE Classic s
All-Cause Mortality (participants affected / at risk) | 0/503
Serious Adverse Events (participants affected / at risk) | 10/503
Other Adverse Events (participants affected / at risk) | 55/503
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | YVOIRE Classic s (N=503)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Extremity injury (Injury, poisoning and procedural complications) | 1
Arrhythmia (Vascular disorders) | 1
Endometrial lesion (Reproductive system and breast disorders) | 1
Gastric polyps (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung cancer (Respiratory, thoracic and mediastinal disorders) | 1
Cervical intraepithelial neoplasia (Reproductive system and breast disorders) | 1
Polyps of duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ectopic pregnancy (Reproductive system and breast disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | YVOIRE Classic s (N=503)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other